CLINICAL TRIAL: NCT06626074
Title: Exploratory Study of MRI Biomarkers of NASH
Acronym: IRM-NASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University Angers (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC23_0262; 2024-A02056-41 (Other: ANSM)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label (Experimental)
  Interventions: Device: Quantitative MRI sequences

INTERVENTIONS:
Device: Quantitative MRI sequences — additional sequences during MRI

SUMMARY:
Metabolic steatosis disease (NAFLD) is a rapidly growing disease in the world, particularly in industrialized countries.

NAFLD is defined by the presence of fatty liver disease. This is a reversible phenomenon that can be estimated by non-invasive means, such as ultrasound. Non-invasive quantification, on the other hand, requires MRI.

Nonalcoholic steatohepatitis (NASH) is the aggressive form of the disease that promotes the accumulation of fibrosis in the liver, which can progress to cirrhosis and its complications.

Currently there is no non-invasive biomarker of NASH and the diagnosis is based solely on liver biopsy.

There is therefore a need for non-invasive biomarkers of NASH in patients with steatosis to diagnose NASH without the use of liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the SNIFF cohort of the Angers hospital where there is a suspicion of NASH requiring a biopsy for which an MRI is requested by a hepatologist as part of the initial assessment of the disease.
* Adult patient
* Free, informed and express (oral) consent of the patient to participate in the study

Exclusion Criteria:

* Contraindication to MRI
* Time between the establishment of the Steatosis/NASH status and the MRI greater than 3 months
* Pregnant, parturient and breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person under compulsion to psychiatric care
* Person subject to a legal protection measure
* Person not affiliated or not covered by a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-09-05 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of new MRI biomarkers for NASH diagnosis | the outcome measurment is performed once during MRI
  NASH is defined by histological criteria

CONTACTS AND LOCATIONS:
Overall Officials: Anita PAISANT, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital, Angers, Angers, France, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).